CLINICAL TRIAL: NCT05294861
Title: Effect of Milk Consumption on Glycemic Control and Gut Microbiome in Type 2 Diabetes
Brief Title: Effect of Milk Consumption on Glycemia and Gut Microbiome in T2D
Acronym: Milk-GM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Prof. Daniela Jakubowicz, MD, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0041-22-WOMC
Record Dates: First submitted 2022-03-13; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Type2Diabetes

STUDY DESIGN:
Intervention Model Description: In a crossover design, the effects of YesMdiet and of NoMdiet on overall glycemia and Gut Microbiome will be assessed in the participants in random order
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YesMdiet (Experimental): After one week baseline, the participants will be assigned to YesMdiet, consuming milk and dairy products for 14 days
  Interventions: Other: YesMdiet
- NoMdiet (Active Comparator): After one week baseline, the participants will be assigned to NoMdiet, consuming another source of protein and without milk or dairy products for 14 days
  Interventions: Other: NoMdiet

INTERVENTIONS:
Other: YesMdiet — In the YesMdiet, participants will consume Milk and Dairy products
  Other Names: Yes Milk diet
  Arms: YesMdiet
Other: NoMdiet — In the YesMdiet, participants will not consume Milk and Dairy products, only other sources of protein
  Other Names: No Milk diet
  Arms: NoMdiet

SUMMARY:
The overall glycemic excursions display circadian variations which are controlled by the circadian clock genes (CCG) and are strongly influenced by meal timing.

Indeed, in T2D, a diet aligned with the CCG, with high-energy and protein breakfast, and reduced in CH dinner (Bdiet) resulted in effective reduction of body weight, HbA1c, and of overall glycemia versus reverse schedule or six meals, with energy and carbohydrates (CH) evenly distributed throughout the day.

in addition to meal timing of Bdiet, the source of protein i.e., Milk and dairy products, by favorable changes in the Guts Microbiome (GM) composition may also play a role in the reduction of overall glycemia of T2D.

The investigators hypothesize that Bdiet schedule with high content of milk and other dairy proteins (YesMdiet), will reduce overall glycemia in T2D, compared to isocaloric and iso-protein Bdiet with another source (nondairy) proteins (NoMdiet).

Study Design: The effect of the two Bdiet interventions on GM will be assessed in T2D participants in a cross-over design, at baseline and after YesMdiet and after NoMdiet, in random order. We expect more favorable changes in glycemic control and in GM composition in YesMdiet versus NoMdiet.

DETAILED DESCRIPTION:
Background: Reduction of the overall glycemic excursion is the main target in the treatment of T2D to reduce HbA1c and cardiovascular risk. The overall glycemic excursions display circadian variations controlled by the circadian clock genes (CG) and are strongly influenced by meal timing.

Indeed, the investigators have recently shown in T2D, that a diet aligned with the CCG, with high-energy and protein breakfast, and reduced in CH dinner (Bdiet) resulted in effective reduction of body weight, HbA1c, and substantial reduction of overall (diurnal and nocturnal) glycemia as compared to the reverse schedule or a diet with six meals, with energy and carbohydrates (CH) evenly distributed throughout the day.

However, in addition to meal timing, the source of protein in Bdiet and the changes of Gut Microbiome (GM) composition, may also play a role in the reduction of overall glycemia. It has been recently shown that consumption of milk and dairy products is associated beneficial effect on overall glycemia. Further, milk and dairy may exert a beneficial effect on overall glycemia by favorable changes in GM composition.

Working hypothesis: Therefore, in this study, we hypothesize that a Bdiet schedule with high content of milk and other dairy proteins (YesMdiet), compared to isocaloric and iso-protein Bdiet with another source (nondairy) proteins (NoMdiet) and may lead to favorable changes in the Gut Microbiota (GM) [Primary end-point] in association with the improvement of overall glycemia in T2D participant under continuous glucose monitoring (CGM) surveillance.

Study Design: The effect of the two Bdiet interventions on GM will be assessed in n=16 participants in a cross-over design, at baseline and after 14 days of Bdiet consuming Milk and dairy products (YesMdiet) or isocaloric Bdiet without milk or dairy products (NoMdiet), in random order in T2D individual undergoing CGM surveillance.

Expected results: We expect more favorable changes in glycemic control and in GM composition in YesMdiet versus NoMdiet.

Scientific Significance: This trial will reveal whether the benefits of Bdiet on glycemic control is further enhanced by milk and dairy consumption, in association with favorable changes in Gut Microbiome

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with T2D < 20 years
* HbA1c ≥ 6.5 %.
* BMI - 28-45 kg/m2
* Men and women 30 -75 years of age inclusive
* Normal liver, kidney, and thyroid functions, and eGFR > 45 mL/min/1.73 m2.
* Type 2 diabetes controlled with diet, lifestyle alone, or with antidiabetics other than insulin (i.e. biguanides, sulfonylureas, glinides, SGLT2 inhibitors, DPP4 inhibitors, GLP-1 analogs), with stable doses for at least 3 months before entering the study.
* Stable weight (less than 5% change in body weight in last 3 months before the study - determined by self-reporting or documentation in clinical records).
* Concomitant medication i.e. antihypertensive, anti-lipidemic, anti-thrombotic drugs will be allowed also on a stable dose for at least 3 months before the beginning of the trial.
* Patients that usually wake up between 06:00 and 08:00 and go to sleep between 22:00 and 24:00.
* Should not have shift work within 6 months of the study and should not have crossed time zones within 2 weeks of the study.
* No change in medication or nutrition supplements or physical activity will be made during the study.

Exclusion Criteria:

* Type 1 diabetes or secondary forms of diabetes.
* Patients with latent autoimmune diabetes in adults (LADA).
* Treatment with insulin.
* Serum creatinine level >2mg/dl. Renal dysfunction: eGFR < 45 mL/min/1.73 m2).
* Hepatic dysfunction: liver disease or transaminase levels > 2.5-fold above normal.
* Major illness with life expectancy < 5 years.
* Malignant neoplasm requiring chemotherapy, surgery, radiation, or palliative therapy within the previous 5 years (with the exception of basal cell skin cancer).
* Those taking psychotropic, anorectic medication, steroid treatment, or illicit drug abuse or alcoholism within one year prior to study onset. Pregnancy or lactation.
* Known hypersensitivity to milk components or lactose intolerance.
* Night or rotating shift workers or those who crossed more than 2 time zones during the 2- week period prior to study onset.
* Not able to give informed consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-28 (Estimated); Primary Completion 2022-10-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome | 14 day
  Gut Microbiome composition will be assessed using 16s rRNA sequencing method after 14 days of YesMdiet

SECONDARY OUTCOMES:
Gut Microbiome | 14 days
  Gut Microbiome composition will be assessed using 16s rRNA sequencing method after 14 days of NoMdiet
Overall Glycemia | 14 days
  Overall Glycemia will be assessed using continuous glucose monitoring CGM during 14 days of either YesMdiet or NoBdiet

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Wolfson Medical Center

IPD SHARING:
Plan to Share IPD: No